CLINICAL TRIAL: NCT07337226
Title: Association of VAgus Nerve Stimulation and Treadmill Training for GAit Rehabilitation in DE Novo Parkinson's Disease (AVANTGARDE-PD)
Brief Title: Association of VAgus Nerve Stimulation and Treadmill Training for GAit Rehabilitation in DE Novo Parkinson's Disease
Acronym: AVANTGARDE-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Massimo Marano, Principal Investigator, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVANTGARDE-PD
Record Dates: First submitted 2025-11-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Parkinson's Disease (PD)
Keywords: Parkinson's disease; Vagus nerve stimulation; non invasive brain stimulation; treadmill training; freezing of gait; rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — salicylhydroxamic acid; 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Exercise Test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- taVNS paired with sensorized treadmill training (STT) and conventional physical therapy (cPT) (Active Comparator): Participants will receive active taVNS, stimulation parameters: 25 Hz frequency, 200 μs pulse width, and intensity adjusted to the individual's sensory threshold, delivered to the left auricular tragus for the duration of each session (~30 minutes). During stimulation, participants will perform treadmill walking on a sensorized treadmill system with simultaneous conventional physical therapy exercises focused on posture, balance, and gait re-education. Sessions will occur three times per week for four weeks (12 sessions total).
  Interventions: Procedure: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS); Other: Conventional Physical Therapy (cPT); Other: Sensorized Treadmill Training (STT)
- taVNS paired with conventional physical therapy (cPT) (Active Comparator): Participants will receive active taVNS (same parameters and device as Arm 1) during conventional physical therapy sessions without treadmill training.
  Sessions will occur three times per week for four weeks.
  Interventions: Procedure: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS); Other: Conventional Physical Therapy (cPT)
- Sham taVNS paired with STT and cPT (Sham Comparator): Sham stimulation will consist of few impulses delivered at 25 Hz for a duration of 60'' before waning, creating the same initial sensation without continuous current delivering.
  Participants will simultaneously undergo treadmill-based and conventional physical therapy as described above.
  Schedule: three sessions per week for four weeks.
  Interventions: Procedure: Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham taVNS); Other: Conventional Physical Therapy (cPT); Other: Sensorized Treadmill Training (STT)
- Sham taVNS paired with cPT (Sham Comparator): Participants will receive sham stimulation (same device and sham procedure as Arm 3) during conventional physical therapy sessions without treadmill training.
  Schedule: three sessions per week for four weeks.
  Interventions: Procedure: Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham taVNS); Other: Conventional Physical Therapy (cPT)

INTERVENTIONS:
Procedure: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Active taVNS delivered at the inner tragus of the left ear (25 Hz, 200 μs, intensity at sensory threshold)
  Other Names: Transcutaneous Auricular Vagus Nerve Stimulation; taVNS; nVNS; tVNS; Transauricular Vagus Nerve Stimulation
  Arms: taVNS paired with conventional physical therapy (cPT); taVNS paired with sensorized treadmill training (STT) and conventional physical therapy (cPT)
Procedure: Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham taVNS) — Sham taVNS using the electrode placement as active taVNS but without electrical stimulation beyond the initial sensation.
  Other Names: Sham transcutaneous auricular vagus nerve stimulation; sham taVNS; sham
  Arms: Sham taVNS paired with STT and cPT; Sham taVNS paired with cPT
Other: Conventional Physical Therapy (cPT) — Conventional Physical Therapy delivered to all groups consist of exercises aimed at posture alignment, reduction of hypertone, balance improvement and overground gait training.
  Other Names: Conventional Physical Therapy; cPT
Other: Sensorized Treadmill Training (STT) — Sensorized Treadmill Training consist of a sensorized gait treadmill training with continuous visual feedback combined with dual cognitive tasks (e.g. repeat digits, repeat sequence of words, counting down the dates).
  Other Names: Sensorized Treadmill Training; STT; treadmill; sensorized treadmill
  Arms: Sham taVNS paired with STT and cPT; taVNS paired with sensorized treadmill training (STT) and conventional physical therapy (cPT)

SUMMARY:
The goal of this clinical trial is to learn if transcutaneous auricular vagus nerve stimulation (taVNS) can improve gait and brain function in people with diagnosis of idiopathic Parkinson's disease (PD) within 6 months. It will also help researchers learn about the safety and biological effects of taVNS when used together with physical therapy.

The main questions it aims to answer are:

* Does taVNS paired with physical therapy improve walking speed and gait performance in people with PD?
* Does taVNS change brain activity or breain perfusion related to movement?
* Does taVNS reduce markers of inflammation and neurodegeneration in blood and saliva? Researchers will compare active taVNS to sham (placebo) stimulation to see if active taVNS works better when paired with physical therapy.

Participants will:

* Attend 12 rehabilitation sessions over 4 weeks (three per week)
* Receive either active or sham taVNS during each session while doing treadmill and conventional physical therapy
* Undergo gait and cognitive testing, MRI scans, and blood and saliva collection before and after treatment
* Return for a follow-up visit four weeks after therapy to check how long the effects last

DETAILED DESCRIPTION:
Parkinson's disease (PD) is characterized by gait disturbance, impaired mobility, and progressive involvement of neural circuits responsible for locomotion and postural control. Although physical therapy is effective, its benefits are often modest and short-lived. Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive neuromodulation technique that activates the auricular branch of the vagus nerve and engages ascending brainstem pathways involved in motor control, arousal regulation, and inflammatory modulation. Previous studies have shown that taVNS can influence subcortical β-band oscillations, improve gait parameters, enhance cognitive performance, and modulate systemic inflammatory markers in individuals with PD.

This randomized, double-blind, sham-controlled clinical trial evaluates whether pairing taVNS with gait-focused rehabilitation enhances motor outcomes and neural plasticity in individuals with de novo PD. Participants are newly diagnosed (≤6 months) and undergo a 4-week rehabilitation program consisting of conventional physiotherapy, with or without sensorized treadmill training. Active or sham taVNS is administered during each therapy session. The study includes four parallel arms to independently assess the contributions of taVNS and treadmill-based gait training.

Outcomes are assessed at baseline (T0), immediately post-intervention (T1), and at a 4-week follow-up visit (T2). Primary and secondary outcomes include quantitative gait parameters, clinical motor scales, cognitive performance, and quality-of-life measures. Exploratory outcomes include changes in cerebral blood flow measured with pseudo-continuous arterial spin labeling (PCASL), functional connectivity during a simulated gait task using fMRI, and blood and salivary biomarkers of inflammation and neurodegeneration (e.g., TNF-α, interleukins, and α-synuclein).

The study aims to determine whether taVNS enhances rehabilitation-induced improvements in gait, whether these benefits persist beyond the treatment period, and whether taVNS induces measurable changes in brain perfusion, functional networks, or circulating biological markers relevant to PD pathophysiology. Results may support the development of a scalable, non-invasive therapeutic approach that can be integrated into early PD management.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD diagnosis within 6 months, confirmed by neurologist specialized in Parkinson's disease and movement disorders;
* Ability to walking independently for at least 10 meters unassisted;
* Age included between 50 and 80;
* MMSE > 24;
* On stable therapy for at least 1 month prior to the experiment.

Exclusion Criteria:

* Clinical and radiological red flags for atypical, vascular parkinsonism or alternative diagnosis (e.g., normal pressure hydrocephalus);
* Levodopa equivalent daily dose > 300 mg;
* Any contraindication for taVNS (e.g., ear lesions, auditory prosthesis)
* Any contraindication for MRI (e.g., non compatible pacemakers or prosthesis, claustrophobic subjects);
* Concomitant neurological, orthopedic or active medical/oncological condition that would affect participating to the study;
* Attempting to other neurorehabilitation programs within 3 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of objective changes in gait speed (m/s) through gait analysis. | Baseline (T0) and Post-intervention (T1, 4 weeks)
  Gait speed (m/s) is measured using a 3D optoelectronic motion-capture system with inertial sensors during level walking on a 10-meter walkway with integrated force platforms. Standard lower-limb reflective markers and surface EMG are used to capture kinematic and muscle-activation patterns. Average gait speed is calculated as the mean forward velocity.

SECONDARY OUTCOMES:
Spatiotemporal and Kinematic Gait Parameters assessment (gait quality parameter). | Baseline (T0), Post-intervention at 4 weeks (T1)
  Spatiotemporal and kinematic gait parameters are measured using a 3D motion-capture system with inertial sensors and surface EMG while participants walk across a walkway with integrated force platforms. Parameters include stance and swing phase duration (s), single and double support time (s), step and stride length (cm) and variability (%), swing speed (m/s) and cadence (steps/min), lower-limb joint flexion-extension angles (°), peak vertical ground reaction force (N/kg), and muscle-activation timing (ms) from surface EMG. All listed parameters will be analyzed collectively as a single composite secondary outcome and will not be reported as separate outcome measures.
Change in Motor Function (MDS-UPDRS Part III Total Score). | Baseline (T0) and Post-intervention at 4 weeks (T1).
  Motor function will be assessed using the Movement Disorder Society Unified Parkinson's Disease Rating Scale, Part III (MDS-UPDRS III), which evaluates bradykinesia, rigidity, tremor, posture, and gait-related motor signs. Total scores range from 0 to 132, with higher scores indicating worse motor impairment. Improvement is reflected by a decrease in the MDS-UPDRS III score.
Cognitive Function (RBANS Total Score) assessment. | Baseline (T0) and Post-intervention at 4 weeks (T1)
  Cognition is assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), which evaluates immediate memory, visuospatial/constructional abilities, language, attention, and delayed memory. Total scores range from 40 (severely impaired) to 160 (very superior), with higher scores indicating better performance.
Quality of Life (PDQ-39 Total and Domain Scores) assessment. | Baseline (T0) and Post-intervention at 4 weeks (T1)
  Quality of life is assessed using the Parkinson's Disease Questionnaire-39 (PDQ-39), which measures mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. Domain and total scores range from 0 to 100, with higher scores indicating poorer quality of life. Improvement is reflected by a decrease in PDQ-39 scores.
Change in Gait Speed from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Average gait speed (m/s) is measured using a 3D motion-capture system during level walking. This outcome represents the change in gait speed between the post-intervention visit (T1) and the follow-up visit (T2) to evaluate persistence of treatment effects.
Change in Spatiotemporal and Kinematic Gait Parameters (gait quality parameter) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Spatiotemporal and kinematic gait parameters (stance and swing duration (s), single and double support time (s), step and stride length (cm) and variability (%), swing speed (cm/s) and cadence (steps/min), joint flexion-extension angles (°), peak vertical ground reaction force (N/kg), and muscle-activation timing (ms)) are assessed with 3D motion capture, force platforms, and surface EMG. All listed parameters will be analyzed collectively as a single composite secondary outcome and will not be reported as separate outcome measures. This outcome reflects change in these parameters from T1 to T2.
Change in Motor Function (MDS-UPDRS Part III Total Score) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Motor function will be assessed using the Movement Disorder Society Unified Parkinson's Disease Rating Scale, Part III (MDS-UPDRS III), which evaluates bradykinesia, rigidity, tremor, posture, and gait-related motor signs. Total scores range from 0 to 132, with higher scores indicating worse motor impairment. Improvement is reflected by a decrease in the MDS-UPDRS III score.
Change in Cognitive Function (RBANS Total Score) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Cognition is assessed with the RBANS, which evaluates immediate memory, visuospatial/constructional abilities, language, attention, and delayed memory. This outcome captures the change in RBANS total score from T1 to T2 to evaluate persistence of cognitive effects. Higher scores indicate better performance.
Change in Quality of Life (PDQ-39) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Quality of life is assessed using the PDQ-39, which measures mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. This outcome represents the change in PDQ-39 total score from T1 to T2, where higher scores indicate poorer quality of life and improvement is reflected by a decrease in scores.
Change in Inflammatory Biomarkers (Serum and Salivary Cytokines) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Serum and salivary levels of inflammatory cytokines (TNF-α, IL-1β, IL-13, IL-10, IL-6) will be measured using standardized ELISA or multiplex immunoassays. Concentrations will be expressed in pg/mL. Cytokines will be analyzed collectively as a composite inflammatory outcome.
Change in Neurodegenerative Biomarker Levels (α-Synuclein) from Post-intervention to Follow-up. | Post-intervention at 4 weeks (T1) and Follow-up at 8 weeks (T2)
  Serum and salivary levels of α-synuclein will be measured using standardized immunoassays. Concentrations will be expressed in ng/mL.

OTHER OUTCOMES:
Imaging Outcomes (PCASL). | Baseline (T0) and Post-treatment at 4 weeks (T1)
  Brain perfusion will be assessed using pseudo-continuous arterial spin labeling (PCASL). Imaging is performed at baseline (T0) and post-treatment (T1). Primary imaging endpoints include:
  - Change in cerebral blood flow (CBF) in locomotor and motor-control regions (PCASL)
Imaging Outcomes (fMRI). | Baseline (T0) and Post-treatment at 4 weeks (T1)
  Functional connectivity will be assessed by functional MRI (fMRI). Imaging is performed at baseline (T0) and post-treatment (T1). The fMRI assessment includes a simulated gait task using a custom pedal system with synchronized visual feedback.
  Primary imaging endpoints include:
  - Change in functional connectivity within gait-related cortical-subcortical networks (fMRI).
Inflammatory Biomarkers (Serum and Salivary Cytokines) | Baseline (T0) and Post-treatment at 4 weeks (T1)
  Serum and salivary levels of inflammatory cytokines (TNF-α, IL-1β, IL-13, IL-10, IL-6) will be measured using standardized ELISA or multiplex immunoassays. Concentrations will be expressed in pg/mL. Cytokines will be analyzed collectively as a composite inflammatory outcome.
Neurodegenerative Biomarker (α-Synuclein) | Baseline (T0) and Post-treatment at 4 weeks (T1)
  Serum and salivary levels of α-synuclein will be measured using standardized immunoassays. Concentrations will be expressed in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Marano, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Campus Bio-Medico, Via Alvaro del Portillo, 200, 00128 Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Not shared due to privacy reasons